CLINICAL TRIAL: NCT04206995
Title: Cancer Sensing: Evaluation of Odour Sampling Techniques to Support the Non-invasive Early Detection of Skin Cancer - Proof of Concept
Brief Title: Cancer Sensing: Evaluation of Odour Sampling Techniques
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Poole Hospital NHS Foundation Trust (Other); Dorset County Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: Skin cancer sensing by VOCs
Record Dates: First submitted 2019-12-13; First posted 2019-12-20 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Solid Phase Microextraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation of odour capturing techniques: To evaluate two odour capturing techniques to compare VOC profiles of cancerous and healthy skin cancer.
  Interventions: Other: Solid Phase Microextraction (SPME); Other: Absorptive patch

INTERVENTIONS:
Other: Solid Phase Microextraction (SPME) — A SPME fibre is held directly above skin cancer, or healthy skin for a period of less than 30 minutes to capture VOCs. No drug will be used. This is to investigate the capability of the technique in capturing VOCs.
Other: Absorptive patch — An adsorptive patch, covering skin cancer and healthy skin sites will be applied for a period of maximum 30 minutes to capture VOCs. No drug will be used. This is to investigate the capability of the technique in capturing VOCs.

SUMMARY:
To evaluate the suitability of two odour capturing techniques for early detection of skin cancer.

DETAILED DESCRIPTION:
The study will investigate the suitability of two odour capturing techniques for early detection of skin cancer. The techniques to capture VOCs are: a) solid phase microextraction (SPME) and b) collection of VOCs via an adsorptive patch, worn on the skin. The objective is to evaluate the suitability of two techniques for collecting VOCs.

Odour samples from cancerous and healthy skin will be captured using the two non-invasive techniques. The techniques will initially be tested in a laboratory environment. They will then be applied in parallel to patients and healthy people. VOC compounds of odour samples will be analysed for their profiles in respect of cancerous and healthy skins. The VOCs profiles will be recorded in a VOC bank for future analysis.

Following the initial tests, patients (n=20) with skin cancer will be recruited from Poole and Dorset County Hospitals. Arrangement will be made to obtain odour samples by positioning patches on the cancerous skin sites (for approximately 30 minutes) of patients and recover them. To obtain samples from healthy people (n=10), staff and students within the university are invited to participate in this research by providing odour samples from their skins using the same type of patches.

In parallel, VOCs from skin cancer patients will also be collected from patients with the SPME fibres described earlier. The SPME device is roughly equivalent in size and shape to a ballpoint pen, from the tip of which an adsorbent fibre can be extended. The SPME device is held statically with a flexible clamp (a weighted clamp which rests on a bench / desk near the patient), and is positioned so that the tip of the fibre rests close to, but not touching, the affected skin area. The fibre needs to be held in place to sample the air above the affected skin for a pre-determined period of time, likely to be 15 - 30 minutes. Specifics such as the sampling time and related factors will be evaluated during the initial laboratory testing. Following the defined time period of sampling, the fibre is retracted into the body of the SPME device (to protect it), and the device is returned to the laboratory for analysis. The high temperatures involved in GCMS analysis cause VOCs captured by the SPME device to be released (desorbed) and they are subsequently swept through the GCMS system for analysis.

The VOC samples from both the techniques will be transported to Bournemouth university for analysis.

The outcome will be the identification of the most suitable VOC collection technique (SPME vs patch) by comparing the VOC profiles of cancerous and healthy skin.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with skin cancer, able to speak and understand written English,
* 18 years or older and
* Capable of giving informed consent.

Exclusion Criteria:

* Patients too weak to speak or give written informed consent;
* Non-English speaking without an interpreter;
* Patients lacking mental capacity to consent, or
* Below the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Skin odour samples are obtained from patients who are diagnosed with cancer and during their visit to Poole or Dorset County Hospitals. Skin odour samples of healthy people will also be obtained from staff and students at Bournemouth University.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Evaluate the suitability of the adsorptive patch for collecting VOCs for analysis for early identification of skin cancer. | 30 minutes
  An adsorptive patch, covering skin cancer and healthy skin sites will be applied for a period of maximum 30 minutes to capture VOCs. No drug will be used. This is to investigate the capability of the technique in capturing VOCs.VOCs for analysis for early identification of skin cancer.
Evaluate the suitability of the Solid Phase Microextraction (SPME) for analysis for early identification of skin cancer. | 30 minutes
  A SPME fibre is held directly above skin cancer, or healthy skin for a period of less than 30 minutes to capture VOCs. No drug will be used. This is to investigate the capability of the technique in capturing VOCs.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Paul, PhD, Study Director — Bournemouth University
Locations (2):
- United Kingdom (2):
  - Dorset County Hospital NHS Foundation Trust, Dorchester, Dorset
  - University Hospitals Dorset NHS Foundation Trust, Poole, Dorset